CLINICAL TRIAL: NCT06038812
Title: Outcome of Non-surgical Periodontal Treatment on Gal-1 & Gal-3 GCF Levels in Periodontitis Patients
Brief Title: Galectin Role in Periodontal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Nayroz Tarrad, associate professor, Fayoum University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: REC-FDBSU/03082023-1/AM
Record Dates: First submitted 2023-08-30; First posted 2023-09-15 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Gingivitis; Periodontitis
MeSH Terms: conditions — Gingivitis; Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Other): patients diagnosed with gingivitis
  Interventions: Diagnostic Test: GCF sample collection
- Group II (Other): patients diagnosed with periodontitis
  Interventions: Diagnostic Test: GCF sample collection; Procedure: non-surgical periodontal treatment
- Group III (Other): healthy control
  Interventions: Diagnostic Test: GCF sample collection

INTERVENTIONS:
Diagnostic Test: GCF sample collection — collecting GCF from deepest sites by paper points
Procedure: non-surgical periodontal treatment — performing scaling and root planning using ultrasonic device and manual curettes
  Arms: Group II

SUMMARY:
This study aimed at exploring the effect of nonsurgical periodontal treatment on galectin 1 and 3 GCF levels in patients having gingivitis, periodontitis stage III compared to periodontally healthy individuals and if galectin-1 and -3 could serve as diagnostic markers and/or therapeutic targets for periodontitis, in addition to revealing their possible role in the periodontal disease.

45 systemically healthy participants were enrolled in this investigation, equally subdivided into three groups of 15 patients each: gingivitis, periodontitis (stage III) and control group with healthy gingiva. Probing depth, clinical attachment level, gingival and plaque index were registered. GCF levels of galectin-1 and -3 were evaluated in all included groups (before and after non-surgical treatment for periodontitis group) using enzyme linked immune-sorbent assay (ELISA) kit.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smokers from both genders.
2. Not suffering from systemic diseases, pregnancy/lactation.
3. Not taking contraceptive pills, antibiotics, anti-inflammatory, or immunosuppressive drugs before inclusion in the study by 6 months.
4. Patients with only gingivitis or periodontitis stage III.
5. Periodontitis patients who did not receive any professional periodontal treatment in the last 6 months.

Exclusion Criteria:

1. smokers.
2. having systemic diseases, pregnancy/lactation.
3. taking contraceptive pills, antibiotics, anti-inflammatory, or immunosuppressive drugs in the past 6 months.
4. Patients having periodontitis any other stage than stage III.
5. Periodontitis patients who receive any professional periodontal treatment in the last 6 months.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
assessment of gal-1 and gal-3 in GCF samples | an average of about 10 months to assess level of gal-1 & -3 after collection of GCF samples at baseline (1st appointment) for all groups and another sample collection after 4 weeks for group II after performing scaling and root planning
  samples are to be sent to biochemistry lab to measure galectin levels

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, Fayoum university, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tarrad NAF, Shaker OG, Elbanna RMH, AbdelKawy M. "Outcome of non-surgical periodontal treatment on Gal-1 and Gal-3 GCF levels in periodontitis patients: a case-control study". Clin Oral Investig. 2024 May 14;28(6):309. doi: 10.1007/s00784-024-05688-1. PMID 38743248